CLINICAL TRIAL: NCT03984006
Title: Early Detection of Autoimmune Thyroid Heart Disease Via Urinary Exosomal Proteins.
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201904095RIND
Record Dates: First submitted 2019-06-04; First posted 2019-06-12 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Thyroid Diseases; Heart Failure
Keywords: Exosome; Urine; Biological marker
MeSH Terms: conditions — Thyroid Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Autoimmune thyroid disease revealed close relationship with heart failure, including the entities of subclinical hyperthyroidism and hypothyroidism. Heart failure is a principal complication of all forms of heart disease. The American College of Cardiology defines HF as a complex clinical syndrome that impairs the ability of the ventricle to fill with or inject blood. In fact, it may be caused by a defect in myocardial contraction, by an impairment in ventricular filling with preserved systolic function ('diastolic HF') or by a combination of both. Earlier detection of probable trend of heart failure in subclinical thyroid diseases is very important in not only Taiwan, Pan-Asia, but all over the aging world. However, it is not currently available.

The investigators will enroll 20 patients with subclinical hyperthyroidism, subclinical hypothyroidism, and collect their urine specimens in outpatient clinic per year.

Prognostic biological markers via this prospective study. The study was designed as prospective pattern, and the investigators will enroll clinical and subclinical thyroid disease with quarterly follow-up, then detect urine exosomal proteins NT-proBNP. The investigators try to find the correlation of outcome with unknown/fresh biomarkers in this study with time-dependent manner.

The investigators hope to find earlier predicting biomarkers for heart dysfunction in autoimmune thyroid disease.

DETAILED DESCRIPTION:
Clinical and subclinical thyroid disease is usually used to describe patients with mild symptoms correlated to hyperthyroid or hypothyroid state. Thyroid ultrasonography could differentiate benign or malignant nodular lesion, together with fine needle aspiration cytology and surgical pathology. Thyrotropin (TSH, thyroid stimulating hormone) is the pivotal investigation in laboratory diagnosis to define subclinical thyroid diseases. An elevated TSH with normal free thyroxine and triiodothyronine levels in serum is defined to be subclinical hypothyroidism, and a subnormal TSH with normal thyroid hormone concentrations to be subclinical hyperthyroidism. Generally, the prevalence of subclinical hypothyroidism and hyperthyroidism were reported as 4% -10% & 1%-2% in general population, respectively. Although subclinical thyroid disease is prevalent, there is still no consensus for screening clinical and subclinical thyroid disease, including hyperthyroidism, hypothyroidism, nodular goiter and thyroid cancer. Under consideration of age, gender or familial history of autoimmune thyroid disease. However, screening for thyroid dysfunction should be considered in some high risk patients, including 1) elderly; 2) history of atrial fibrillation; 3) previous thyroid disease history; 4) other confirmed autoimmune diseases; 5) neck exposure of radiation (for example, nasopharyngeal cancer, post-radiation); 6) family history of probable autoimmune thyroid disease, and 7) pregnant state with prior thyroid disease history. Therapeutic decision for clinical and subclinical thyroid dysfunction should be considered individually. Therapeutic options will be anti-thyroid medications and/or radioactive iodine, and thyroidectomy could be considered with larger goiters for hyperthyroidism. For clinical and subclinical hypothyroidism, the therapeutic consideration should be aimed on reduction of progression to overt hypothyroidism, improving heart function, correction of dyslipidemia, and relieving senescence depressive mood. Thyroid ultrasonography will help us to keep long term observation of thyroid structural change. But long term outcome for treatment of such functional and structural thyroid diseases had not been recorded delicately in Taiwan. Further investigations should be observed in the future. The investigators hope to check the relationship between various thyroid diseases and biochemical survey/ultrasonography. The purpose of this study is aiming for early prevention and detection the potential risk factors for thyroid diseases in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed patients with autoimmune thyroid disease (subclinical hyperthyroidism, subclinical hypothyroidism)

Exclusion Criteria:

* Unclearly diagnosed patients with autoimmune thyroid disease (subclinical hyperthyroidism, subclinical hypothyroidism)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will enroll 20 patients with subclinical hyperthyroidism, subclinical hypothyroidism, and collect their urine specimens in outpatient clinic per year.
  The investigators will analyze the urine exosomal proteins and probable biological markers, including NT-proBNP and other proteins.
  The investigators hope to find the prognostic biological markers via this prospective study. The investigators further hope to find newly therapeutic and follow-up pathway for such patients with autoimmune thyroid disease (subclinical hyperthyroidism, subclinical hypothyroidism).
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Change of serum thyroglobulin level | Within 12 months
  Comparison to enrollment or between 2 groups
Change of serum free T4 level | Within 12 months
  Comparison to enrollment or between 2 groups
Change of serum TSH level | Within 12 months
  Comparison to enrollment or between 2 groups
Change of anti-thyroglobulin level | Within 12 months
  Comparison to enrollment or between 2 groups
Urinary exosomal NT-proBNP detection | Within 12 months
  Comparison to enrollment or between 2 groups
2-D Cardiac Doppler ultrasonography evaluation | Within 12 months
  Comparison to enrollment or between 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: CHIH-YUAN WANG, Doctor, Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No